CLINICAL TRIAL: NCT05709106
Title: A Prospective Real World Study of Rimegepant in the Treatment of Migraine
Status: Completed | Type: Observational
Sponsor: Ruijin-Hainan Hospital Shanghai Jiao Tong University School Of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: ky2022005
Record Dates: First submitted 2023-01-13; First posted 2023-02-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — rimegepant sulfate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rimegepant treatment group: this group would use Rimegepant 75mg ODT, use it when needed for 1year
  Interventions: Drug: Rimegepant 75 MG

INTERVENTIONS:
Drug: Rimegepant 75 MG — Migraine patients would take Rimegepant 75 MG to treat or prevent a migraine attack and patients would be followed up for 1 year

SUMMARY:
The goal of this observational study is to test the effectiveness and safety of Rimegepant in the treatment of migraine patients in real world.

The main questions it aims to answer are:

* [question 1] the effectiveness and safety of Rimegepant in the acute treatment of migraine
* [question 2] the effectiveness and safety of Rimegepant in the long-term treatment of migraine.

  1. Participants will be asked to take Rimegepant when they need to treat or prevent a migraine attack.
  2. Participants will be asked to record the efficacy data at 0.5, 1, 2, 24, 48h post dose and report any AE to evaluate the effectiveness and safety of Rimegepant in the acute treatment of migraine
  3. Participants will be asked to track monthly migraine days and the use of Rimegepant, finish 2 PROs during the follow-ups, report any AE to evaluate the effectiveness and safety of Rimegepant in the long-term treatment of migraine.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed as migraines (with or without aura) consistent with a diagnosis according to the International Classification of Headache Disorders, 3rd Edition, beta version
* Rimegepant is prescribed by the physician for the treatment of patients with migraine.
* Patients signed written informed consent.
* Male and Female subjects ≥ 18 years and older
* Patients is not participated in other concurrent interventional clinical studies.

Exclusion Criteria:

* The patients with severe visual, hearing, language, intelligence, memory, and consciousness disorders, are unable to cooperate with the completion of the questionnaire and follow-up.
* Pregnant patients
* Lactating female patients
* Patients who are highly dependent on medical care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted in the headache clinic of Ruijin-hainan hospital. Participants meeting the inclusion and exclusion criteria will be enrolled continuously.
Sampling Method: Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2024-10-06 (Actual); Study Completion 2025-04-09 (Actual)

PRIMARY OUTCOMES:
Change From Baseline on the percentage of participants that are pain relief at 2 hours post-dose during the migraine attack | Difference between baseline and 2 hours post-dose of Rimegepant
  Pain Relief at 2 hours post-dose will be assessed using the number of subjects that report a pain level of moderate or severe at baseline and then report a pain level of none or mild at two hours post-dose.

SECONDARY OUTCOMES:
Change From Baseline on percentage of participants that are pain relief at 0.5,1,24 and 48 hours post-dose during the migraine attack | Difference between baseline and 0.5, 1, 24 and 48 hours post-dose of Rimegepant
  Pain Relief at 0.5,1,24 and 48 hours post-dose will be assessed using the number of subjects that report a pain level of moderate or severe at baseline and then report a pain level of none or mild at 0.5,1,24 and 48 hours post-dose.
Change From Baseline on the percentage of subjects able to function normally, at 0.5, 1, 2, 24 and 48 hours post-dose, will be accessed by the Functional Disability scale | Difference between baseline and 0.5, 1, 2, 24 and 48 hours post-dose of Rimegepant
  The ability to function normally will be measured using the number of subjects that self-report as "normal" on the Functional Disability scale
Change From Baseline on the percentage of participants that are pain freedom at 0.5,1, 2, 24 and 48 hours post-dose during the migraine attack | Difference between baseline and 0.5, 1, 2, 24 and 48 hours post-dose of Rimegepant
  Pain freedom will be assessed using the number of evaluable subjects that report no pain at 0.5,1,2,24 and 48 hours post-dose. Pain will be measured on a 4 point Likert scale (0=none, 1=mild, 2=moderate, 3=severe).
Change From Baseline on the percentage of participants that are freedom from Most Bothersome Symptoms MBS (nausea, phonophobia or photophobia) at 0.5,1,2,24 and 48 hours post-dose during the migraine attack | Difference between baseline and 0.5, 1, 2, 24 and 48 hours post-dose of Rimegepant
  Freedom from Most Bothersome Symptom will be measured using the number of subjects that report the absence of their MBS (nausea, phonophobia or photophobia) and will measured as (0=absent, 1=present)
Change From Baseline in the Mean Number of Migraine Days Per Month Over the 12 months follow-up period. | From baseline to 12 months follow-up period
  A migraine day: any calendar day in which the participant experienced a qualified migraine headache (onset, continuation, or recurrence of the migraine headache). If the participant took a migraine-specific medication during aura or to treat headache on a calendar day, it was counted as a migraine day regardless of the duration and pain features/associated symptoms. (A month is defined as 4 weeks for the purpose of this protocol).The change from baseline was calculated as the number of monthly migraine days during the every 4 weeks of the 12 months follow-up period minus number of monthly migraine days of baseline.Baseline is defined as the number of migraine days during the last 28 days prior to the recruiting date.
Change from baseline in the Migraine-Specific Quality-of-Life Questionnaire v 2.1 (MSQ) total score and Headache Impact Test (HIT-6) total score at month 3,6,12 in the 12 months follow-up | From baseline and month 3,6,12 in the 12 months follow-up
  The MSQ v2.1 is a 14-item questionnaire designed to measure health-related quality of life impairments attributed to migraine in the past 4 weeks.The HIT-6 is a 6-question assessment used to measure the impact headaches have on a participant's ability to function on the job, at school, at home, and in social situations.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Liu, Principal Investigator — Ruijin-Hainan Hospital Shanghai Jiao Tong University School Of Medicine
Locations (1):
- Ruijin-Hainan Hospital Shanghai Jiao Tong University School of Medicine, Boao, Hainan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yang Z, Wang X, Niu M, Wei Q, Zhong H, Li X, Yuan W, Xu W, Zhu S, Yu S, Liu J, Yan J, Kang W, Huang P. First real-world study on the effectiveness and tolerability of rimegepant for acute migraine therapy in Chinese patients. J Headache Pain. 2024 Sep 27;25(1):160. doi: 10.1186/s10194-024-01873-5. PMID 39333875